CLINICAL TRIAL: NCT04836273
Title: Ready-to-use Dasiglucagon for the Treatment of Postprandial Hypoglycaemia in Roux-en-Y Gastric Bypass Operated Patients
Brief Title: Treatment of Post-bariatric Hypoglycaemia
Acronym: SHERRY
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Filip Krag Knop (Other)
Collaborators: Zealand Pharma (Industry)
Responsible Party: Sponsor-Investigator, Filip Krag Knop, Principal Investigator, Clinical Professor, University Hospital, Gentofte, Copenhagen
Organization: University Hospital, Gentofte, Copenhagen (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CKN-DASI120-RYGB; 2020-005241-16 (EudraCT Number)
Record Dates: First submitted 2021-03-26; First posted 2021-04-08 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-02

CONDITIONS: Hyperinsulinemic Hypoglycemia; Postprandial Hypoglycemia
MeSH Terms: conditions — Congenital Hyperinsulinism; Hypoglycemia | interventions — dasiglucagon

STUDY DESIGN:
Intervention Model Description: 4 weeks x 4 weeks with an interposed washout period of 1 week
Who Masked: Participant, Investigator
Masking Description: Double-blind (participants and investigator)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 120 µg dasiglucagon (Experimental): Subcutaneous 120 µg dasiglucagon self-administration
  Interventions: Drug: Dasiglucagon; Device: HyoPen
- Placebo (Placebo Comparator): Subcutaneous placebo self-administration
  Interventions: Device: HyoPen; Drug: Placebo

INTERVENTIONS:
Drug: Dasiglucagon — Abdominal s.c. self-administration 120 µg of dasiglucagon when blood glucose levels are below 3.9 mmol/L or interstitial glucose levels below 3.5 mmol/L. The frequency of the intervention is approximately once a day.
  Other Names: ZP4207
  Arms: 120 µg dasiglucagon
Device: HyoPen — multi-dose reusable pen injector
  Other Names: Zealand Pen
Drug: Placebo — Abdominal s.c. self-administration with placebo when blood glucose levels are below 3.9 mmol/L or interstitial glucose levels below 3.5 mmol/L. The frequency of the intervention is approximately once a day.
  Arms: Placebo

SUMMARY:
This is an investigator-initiated, proof-of-concept, randomised, double-blind, placebo-controlled, single-centre phase II study aiming to evaluate the efficacy, safety and tolerability of self-administered subcutaneous 120 µg dasiglucagon with an investigational trial device (i.e. a multi-dose reusable pen) for the treatment of postprandial hypoglycaemia after Roux-en-Y gastric bypass (RYGB) surgery. The study is divided into an in-patient and out-patient part.

The primary aim of the study is to compare the effects of self-administered 120 µg dasiglucagon versus placebo on continuous glucose monitoring (CGM)-assessed time spent in hypoglycaemia in RYGB-operated individuals in an out-patient setting.

DETAILED DESCRIPTION:
Study design:

Before inclusion in the study, the participants will complete a screening visit and a blinded 14-day continuous glucose monitoring (CGM) run-in period to ascertain a regular occurrence of postprandial hypoglycaemia (IG <3.9 mmol/l, ≥3 times/week). After enrolment in the study, the participants will wear a CGM for the entirety of the study period (apart from the four weeks before the follow-up visit). Prior to the first mixed meal test (MMT) during the in-patient part, the subjects will be randomised into one of four double-blinded treatment sequences consisting of an in-patient part (two MMTs) follow by a nine weeks out-patient part (two times four weeks per out-patient part with an interposed washout period of one week) and ended with a follow-up visit four weeks after out-patient part completion.

During the in-patient part, the participants will undergo two separate MMTs, with a minimum of 7 days in-between, accompanied by one of the following double-blind, randomised, placebo-controlled crossover interventions:

1. Subcutaneous placebo self-administration
2. Subcutaneous 120 µg dasiglucagon self-administration

The out-patient part is divided into two double-blinded, randomised, placebo-controlled crossover out-patient parts with of the following interventions:

1. Subcutaneous placebo self-administration
2. Subcutaneous 120 µg dasiglucagon self-administration

ELIGIBILITY:
Inclusion Criteria:

* Documented postprandial hypoglycaemia (IG <3.9 mmol/l, ≥3 times/week) assessed by 14-days of blinded CGM recording
* Haemoglobin levels for women >7.3 mmol/l and for men >8.3 mmol/l
* Ferritin >10 μg/l
* Cobalamin >150 pmol/l
* Fasting plasma glucose concentration within the range of 4.0-6.0 mmol/l
* Normal electrocardiogram (ECG)
* Negative urine human chorionic gonadotropin (hCG) (for fertile women)

Exclusion Criteria:

* Treatment with medication(s) affecting insulin secretion, glucose metabolism or any antidiabetic drugs
* Treatment with antipsychotics
* Current participation in another clinical trial with administration of investigational drug
* Previous exposure to dasiglucagon (also known as ZP4207) within the last 30 days prior screening
* History of liver disease that is expected to interfere with the anti-hypoglycaemic action of glucagon (e.g. liver failure or cirrhosis)
* Pregnancy
* Breastfeeding
* Major surgery within 30 days before screening
* Alcohol abuse (per investigator assessment)
* Any factors that, in the opinion of the site principal investigator or clinical protocol chair, would interfere with the safe completion of the study, including medical conditions that may require hospitalization during the trial
* History of pheochromocytoma or insulinoma
* History of hypersensitivity or allergic reaction to dasiglucagon or any of the excipients
* Known or suspected allergies to glucagon or related products

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-08-20 (Actual); Primary Completion 2022-05-15 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Time spent in hypoglycaemia (IG < 3.9 mmol) | During the four weeks of placebo and dasiglucagon treatment.
  The primary endpoint is the percentage of time in hypoglycaemia (IG <3.9 mmol/l) assessed by CGM during the out-patient part.

SECONDARY OUTCOMES:
Time (percent or minutes) spent in serious hypoglycaemia (IG <3.0 mmol/l) | During the four weeks of placebo and dasiglucagon treatment.
Frequency of hypoglycaemic events (IG <3.9 mmol/l and <3.0 mmol/l, respectively) | During the four weeks of placebo and dasiglucagon treatment.
Glycaemic time in range defined as: 1) hypoglycaemia (<3.9 mmol/l), 2) normoglycaemia (3.9-10.0 mmol/l), and 3) hyperglycaemia (>10.0 mmol/l) | During the four weeks of placebo and dasiglucagon treatment.
Frequency of hyperglycaemic events (IG >7.8 mmol/l and >10.0 mmol/l, respectively) | During the four weeks of placebo and dasiglucagon treatment.
Glycaemic variability assessed as coefficient of variance (CV) | During the four weeks of placebo and dasiglucagon treatment.
Glycaemic variability assessed as standard deviation (SD) | During the four weeks of placebo and dasiglucagon treatment.
Recovery of BG 15 minutes after trial drug administration (as measured by finger prick (BG >3.9 mmol/l)) | During the four weeks of placebo and dasiglucagon treatment.
Change in QoL as assessed by the World Health Organization's quality of life assessment (WHOQOL-BREF) | During the four weeks of placebo and dasiglucagon treatment.
  likert scale, zero (very poor) to five (very good)
Change in hypoglycaemic symptoms will be evaluated by Edinburgh Hypoglycaemia Symptom Scale (EHSS) | During the four weeks of placebo and dasiglucagon treatment.
  likert scale, zero (not a all) to seven (a lot)
Change in fear of hypoglycaemia as assessed by Hypoglycaemia Fear Scale (HFS-II) | During the four weeks of placebo and dasiglucagon treatment.
  likert scale, zero (never) to four (always)
Change in administration frequency (as measured by percentage) | During the four weeks of placebo and dasiglucagon treatment.
Nadir plasma glucose as assessed both as 1) absolute lowest value, and 2) a mean of three consecutive glucose measurements during the 240-minute MMT | Two hundred forty minutes of mixed meal test
  Nadir plasma glucose after the postprandial peak during the MMT in the in-patient part
Recovery of BG 15 minutes after administration (as measured by finger prick (BG >3.9 mmol/l)) | Two hundred forty minutes of mixed meal test
  After the postprandial peak during the MMT in the in-patient part
Time spent in level 1 and level 2 hypoglycaemia (<3.9 and <3.0 mmol/l, respectively) from study drug administration until 240 minutes | Two hundred forty minutes of mixed meal test
  After the postprandial peak during the MMT in the in-patient part
Glycaemic rescue intervention due to critically low plasma glucose concentration (<1.8 mmol/l) | Two hundred forty minutes of mixed meal test
  During the MMT in the in-patient part
Time spent in hyperglycaemia (>7.8 mmol/l) from study drug administration until 240 minutes | Two hundred forty minutes of mixed meal test
  During the MMT in the in-patient part
Peak plasma glucose concentration after study drug administration | Two hundred forty minutes of mixed meal test
  During the MMT in the in-patient part
Counter-regulatory hormonal response | Two hundred forty minutes of mixed meal test
  Measured as area under the curve (AUC) and / or incremental (iAUC) as appropriate, peak values and values at nadir plasma glucose concentration during the MMT in the in-patient part. glucagon-like peptide 1 (GLP-1), glucagon-like peptide 2 (GLP-2), glucose-dependent insulinotropic polypeptide (GIP)
Changes in blood pressure | Two hundred forty minutes of mixed meal test
  During the MMT in the in-patient part
Changes in heart rate | Two hundred forty minutes of mixed meal test
  During the MMT in the in-patient part
Frequency and severity of adverse events (AE)s and serious adverse events (SAE)s from signed consent form to end of study (visit 4 / follow-up visit) | Through study completion which is an average of 16 weeks
  Safety endpoint
Frequency and severity of adverse events (AE)s and serious adverse events (SAE)s during the in-patient part MMTs | During the in-patient part (MMTs) 0-240 minutes / Two hundred forty minutes of mixed meal test
  Safety endpoint
Percentage (%) of participants with treatment-induced or treatment-boosted anti-dasiglucagon antibodies who did not have anti-dasiglucagon antibodies at baseline | Through study completion which is an average of 16 weeks
  Safety endpoint
Device failures/ malfunctions occurring during the trial. | Through study completion which is an average of 16 weeks
  Device endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Filip K Knop, MD, PhD, Principal Investigator — Center for Clinical Metabolic Research at Gentofte Hospital
Locations (1):
- Center for Clinical Metabolic Research, Herlev-Gentofte Hospital, Hellerup, Denmark

IPD SHARING:
Plan to Share IPD: No